CLINICAL TRIAL: NCT06097390
Title: A Study Investigating the Pharmacokinetic Properties When Dosing Different Formulations of Semaglutide to Healthy Male Participants - Oral Formulation III
Brief Title: A Research Study Looking at New Protein-based Tablets in Healthy Men - Oral Formulation III
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9501-4924; U1111-1289-1040 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Healthy Participants
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1: Semaglutide J then Semaglutide K (Experimental): Oral semaglutide J will be administered in treatment period 1 followed by semaglutide K in treatment period 2.
  Interventions: Drug: Semaglutide
- Sequence 2: Semagultide K then Semaglutide J (Experimental): Oral semaglutide K will be administered in treatment period 1 followed by semaglutide J in treatment period 2.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Oral administration

SUMMARY:
In this study, a known medicine called 'semaglutide' will be tested in two different tablet versions. The two tablets differ in the way these have been manufactured. The aim of the study is to investigate the amount of active ingredient in the blood after dosing the different tablet versions. Participants will receive one tablet version for 10 days (first treatment period) and the other version for 10 days (second treatment period). The treatment arm participants will be assigned to is decided by chance. The study will last for about 23 weeks for each participant. The study will enroll healthy male participants.

ELIGIBILITY:
Key inclusion criteria:

* Body mass index (BMI) between 22.0 and 31.9 kilograms per meter square (kg/m^2) (both inclusive) at screening.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Key exclusion criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Any disorder which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Use of prescription medicinal products or non-prescription drugs, except routine vitamins, topical medication not reaching the systemic circulation and occasional use of paracetamol (acetaminophen) and ibuprofen, within 14 days before screening.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Adjusted AUC0-24h,sema; adjusted area under the semaglutide plasma concentration-time curve | From 0 to 24 hours after dosing on day 80 and 90
  Measured in hour*nanomoles per liter (h*nmol/L).

SECONDARY OUTCOMES:
Adjusted Cmax,0-24h,sema; adjusted maximum observed semaglutide plasma concentration | From 0 to 24 hours after dosing on day 80 and 90
  Measured in nanomoles per liter (nmol/L).
Adjusted tmax,0-24h,sema; time to adjusted maximum observed semaglutide plasma concentration | From 0 to 24 hours after dosing on day 80 and 90
  Measured in hours.
t½,sema; the terminal half-life of semaglutide | From 0 to 840 hours after dosing on day 90
  Measured in hours.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Altasciences Clinical Company, Inc, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com